CLINICAL TRIAL: NCT05505734
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Event-driven, Decentralized, Phase IIIb Study Comparing PT027 With PT007 Administered as Needed in Participants 12 Years of Age and Older With Asthma (BATURA)
Brief Title: A Comparison of PT027 vs PT007 Used as Needed in Participants With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV007
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Metered-dose inhaler (MDI); Leukotriene receptor agonist (LTRA); Inhaled corticosteroid (ICS); Short -acting β2agonist (SABA)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PT027 (Experimental): Participants will receive Budesonide and Albuterol Sulfate Pressurised Inhalation Suspension 160/180 μg up to a maximum of 12 inhalations to max dose.
  Interventions: Drug: BDA MDI
- PT007 (Experimental): Participants will receive Albuterol Sulfate Pressurised Inhalation Suspension 180 μg up to a maximum of 12 inhalations to max dose.
  Interventions: Drug: AS MDI

INTERVENTIONS:
Drug: BDA MDI — Participants will receive Budesonide and Albuterol Sulfate MDI 80/90 μg per Actuation 1 to 6 doses (2 inhalations/dose) per day as needed via Oral inhalation route.
  Arms: PT027
Drug: AS MDI — Participants will receive Albuterol Sulfate MDI 90 μg per Actuation 1 to 6 doses (2 inhalations/dose) per day as needed via Oral inhalation route.
  Arms: PT007

SUMMARY:
This is a US study comparing the efficacy and safety of BDA MDI [Budesonide/Albuterol Sulfate (BDA) metered dose inhaler (MDI)] with AS [Albuterol Sulfate] MDI, both are administered as needed for up to 12 months.

DETAILED DESCRIPTION:
This is a phase IIIb, multicenter, randomized, double-blind, parallel-group, event-driven, variable-length, decentralized study.

Participants from around 40 to 50 centers located in the US will be screened and randomized 1:1 to receive one of the following two treatments to be used as needed: BDA MDI (160/180 μg) and AS MDI (180 μg). Participants 12 years of age and older with asthma will be recruited with all visits conducted virtually.

Eligible participants must be using as-needed SABA (Short -acting β2agonist) alone, or as-needed SABA on a background of either low-dose ICS (Inhaled corticosteroid) or a LTRA (Leukotriene receptor agonist), for the treatment of asthma.

Participants will be stratified by pre-study asthma medication (SABA only, low-dose ICS + SABA and LTRA + SABA) and number of prior severe exacerbations (0, ≥1) in the 12 months prior to the Screening visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥12 years of age, at the time of signing the electronic informed consent form (eICF). For participants from 12 years of age to age of majority, their parents/legal guardian must provide signed consent, as appropriate, and participants will sign an assent form.
2. Diagnosis of asthma by a prescribing healthcare professional. Protocol-specified documentation of asthma diagnosis is required to confirm diagnosis of asthma.
3. Participants actively using SABA alone or SABA on a background of either low-dose ICS or LTRA.
4. Self-reported use of a SABA on ≥2 occasions, in response to symptoms (ie, not for exercise prophylaxis only), in the previous 2 weeks prior to enrollment.
5. An Asthma Impairment and Risk Questionnaire (AIRQ) score of ≥2 at Screening (Visit1/re-screen) and Randomisation (Randomization (Visit2) where applicable. Note, where screening Visit1/re-screen and randomization occur on the same day, AIRQ will only be completed once.
6. Females of child-bearing potential must have a negative pregnancy test prior to randomization and agree to use an acceptable method of contraception throughout the study.
7. Male participants who are in heterosexual relationships must be surgically sterile or agree to use an effective method of contraception (condom) if the female partner does not use contraception from the date the eICF is signed until 2 weeks after their last dose.

Exclusion Criteria:

1. Any evidence of significant lung disease other than asthma, such as chronic obstructive pulmonary disease, emphysema, idiopathic pulmonary fibrosis, sarcoidosis etc or any other significant disease (like malignancies or severe chronic diseases) that by Investigator judgment would interfere with the participant being able to comply with study procedures or complete the study.
2. Hospitalization due to asthma in the 3 months prior to enrollment or self-reported admission to the Intensive Care Unit with life-threatening asthma at any time in the past
3. Self-reported use of inhaled Long-Acting Beta-Agonists (LABA), theophylline, inhaled anticholinergic agent, cromone or medium/high dose ICS daily, as regular maintenance asthma therapy in the 3 months prior to enrollment
4. Self-reported use of systemic corticosteroids (SCS) for the treatment of asthma and any other condition in the 6 weeks prior to enrollment
5. Participants with a home supply of oral corticosteroids (OCS) to be used in the case of an asthma exacerbation or any other condition that could require a course of OCS, who are not willing to commit to the treating physician to stop using this medication for the duration of the study.
6. Receipt of any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab, tezepelumab) or investigational biologic for the treatment of asthma at any time in the past
7. Receipt of bronchothermoplasty
8. Use of a SABA prophylactically primarily to prevent exercise induced bronchospasm (EIB) and not to treat symptoms
9. Currently receiving systemic treatment with potent cytochrome P3A4 inhibitors (eg, ketoconazole, itraconazole, and ritonavir)
10. Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
11. Previous screening, enrollment or randomization in the present study.
12. For females only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
13. Participants without access to a smartphone or the internet.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2516 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig LaForce, MD, Principal Investigator — North Carolina Clinical Research
Locations (53):
- United States (53):
  - Pulmonary Associates of Mobile PC, Mobile, Alabama
  - One of a Kind Clinical Research Center, Paradise Valley, Arizona
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Kern Research Inc., Bakersfield, California
  - Science 37, Culver City, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Allergy & Asthma Medical Group and Research (AAMGRC) - Allergy, Asthma and Immunology, San Diego, California
  - Clinical Research of California, Walnut Creek, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - Velocity Clinical Research, Denver, Denver, Colorado
  - Helix Biomedics, Boynton Beach, Florida
  - Allergy and Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - Centricity Research, Columbus, Georgia
  - Lifeline Primary Care, Lilburn, Georgia
  - Javara Inc./Privia Medical Group Georgia, LLC, Savannah, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research, Lafayette, Louisiana
  - Javara Inc., Annapolis, Maryland
  - Baltimore Early Phase Clinical Unit (EPCU), Baltimore, Maryland
  - Chesapeake Clinical Research, White Marsh, Maryland
  - Genesis Clinical Research and Consulting, LLC, Fall River, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Mankato Clinic, Mankato, Minnesota
  - Spectrum Clinical Research, Kansas City, Missouri
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Midwest Regional Health Services, LLC/CCT Research, Omaha, Nebraska
  - Meridian Clinical Research, Endwell, New York
  - Modern Migraine MD/CTNX, New York, New York
  - Javara Inc., Charlotte, North Carolina
  - Javara Inc/Wake Forest Health Network, LLC, Clemmons, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wilmington Health (Innovo Research), Wilmington, North Carolina
  - Buckeye Health and Research, Columbus, Ohio
  - Velocity Clinical Resarch - Medford, Medford, Oregon
  - Northwest Research Center, Portland, Oregon
  - Hatboro Medical Associates, Hatboro, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - CVS Health, Woonsocket, Rhode Island
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - Velocity Clinical Research, Greenville, Greenville, South Carolina
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - Privia Medical Group Gulf Coast, Cypress, Texas
  - CardioVoyage LLC, Denison, Texas
  - Texas Health Care, PLLC d/b/a Privia Medical Group- North Texas, Fort Worth, Texas
  - Allure Health at Mt Olympus Medical Research, Friendswood, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Mt. Olympus Medical Research, Sugar Land, Texas
  - South Ogden Family Medicine clinic, Ogden, Utah
  - Velocity Clinical Research -Salt Lake City, West Jordan, Utah
  - Meridian Clinical Research, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LaForce C, Albers F, Danilewicz A, Jeynes-Ellis A, Kraft M, Panettieri RA Jr, Rees R, Bardsley S, Dunsire L, Harrison T, Sobande O, Surujbally R, Trudo F, Cappelletti C, Papi A, Beasley R, Chipps BE, Israel E, Pandya H, Clancy M, Bacharier LB; BATURA Investigators. As-Needed Albuterol-Budesonide in Mild Asthma. N Engl J Med. 2025 Jul 10;393(2):113-124. doi: 10.1056/NEJMoa2504544. Epub 2025 May 19. PMID 40388330
- See also: Study Design Publication — http://pubmed.ncbi.nlm.nih.gov/39193207/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was screened on 2 September 2022. Participants were enrolled at 54 sites in the United States. Primary and first secondary objectives were tested at the interim analysis, on data collected up to 22 April 2024. Following the decision to stop the study early for overwhelming efficacy, participants were instructed to attend their end of study visits. The last participant last visit occurred on 22 August 2024 and final database lock was achieved on 20 September 2024.
Pre-assignment Details: A total of 5,221 participants were screened for this study, of which 2,516 participants were randomized to treatment; 2,705 were ineligible for participation in the trial. Of the 2,516 participants randomized, the full analysis set (ages 12 years and above) comprised of 2,421 participants as 95 participants discontinued the study prior to dosing randomized treatment.
Groups:
- BDA MDI (PT027) 160/180 μg: Budesonide/albuterol sulfate, BDA MDI, PT027
  Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg: Budesonide/albuterol sulfate combination inhalation aerosol
- AS MDI (PT007) 180 µg: Albuterol sulfate MDI, PT007
  Albuterol sulfate metered-dose inhaler 180 μg: Albuterol sulfate inhalation aerosol
Period: Overall Study
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Started | 1257 | 1259
Full Analysis Set; >=12 Years | 1209 | 1212
Full Analysis Set; >=18 Years | 1180 | 1173
Completed | 903 | 894
Not Completed | 354 | 365
Not completed — Withdrawal by Subject | 51 | 64
Not completed — Adverse Event | 6 | 20
Not completed — Protocol Violation | 8 | 15
Not completed — Lack of therapeutic response | 0 | 1
Not completed — Lost to Follow-up | 247 | 237
Not completed — Physician Decision | 22 | 13
Not completed — Death | 2 | 1
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Other | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg | Total
Number analyzed (Participants) | 1209 | 1212 | 2421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 39 | 68
  Between 18 and 65 years | 1100 | 1073 | 2173
  >=65 years | 80 | 100 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (14.33) | 42.9 (14.68) | 42.7 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 810 | 843 | 1653
  Male | 399 | 369 | 768
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 156 | 136 | 292
  Not Hispanic or Latino | 1052 | 1075 | 2127
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 848 | 849 | 1697
  Black or African American | 219 | 219 | 438
  Asian | 28 | 28 | 56
  Native Hawaiian or other Pacific Islander | 2 | 2 | 4
  American Indian or Alaska Native | 9 | 5 | 14
  Multiple | 19 | 24 | 43
  Other | 47 | 52 | 99
  Not Reported | 37 | 32 | 69
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to First Severe Asthma Exacerbation, While on Treatment Strategy, Interim Analysis Data Cut-off (Participants Aged >=12 Years)
Description: The time to first severe asthma exacerbation was analyzed under the While on Treatment strategy in the Full analysis set (FAS) and was defined as the length in days from treatment initiation until the date of the first severe asthma exacerbation event. Participants were censored at treatment discontinuation, a step-up in maintenance therapy, or interim analysis DCO. An asthma exacerbation was considered severe if it resulted in at least one of the following: use of systemic steroids for at least 3 days, inpatient hospitalization due to asthma or emergency room visit that required systemic steroids, or death due to asthma. The primary outcome measure was analyzed at the interim analysis (22 April 2024). Since the primary objective was met at the interim analysis, it was not re-tested at final database lock. Since fewer than 50% of participants had an exacerbation event, the median survival time could not be calculated and instead the number of participants with an event is reported.
Time Frame: From treatment initiation until the earliest occurrence of study completion, treatment discontinuation, step-up in maintenance therapy, or interim analysis DCO, up to one year following treatment initiation.
Population: Full analysis set; >=12 years
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1209 | 1212
Participants | 62 | 110
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Hazard ratios, 95% confidence intervals for hazard ratios and p-values are estimated using a Cox regression model with treatment group, pre-study asthma therapy, and number of severe exacerbations in the last 12 months prior to randomization as factors. A hazard ratio less than 1 favors the BDA MDI treatment group; Test type: Superiority; p < 0.001, Regression, Cox — The pre-specified alpha (type I error) at the IA was set at 0.003 for the primary and first secondary endpoint; Hazard Ratio (HR) = 0.535, 95% CI 2-sided [0.392 to 0.730]

2. Secondary Outcome: Time to First Severe Asthma Exacerbation, Treatment Policy Strategy, Interim Analysis Data Cut-off (Participants Aged >=12 Years)
Description: The time to first severe asthma exacerbation was analyzed under the Treatment Policy strategy in the Full analysis set (FAS) and was defined as the length in days from treatment initiation until the date of first severe asthma exacerbation occurred. Participants were censored at study completion or withdrawal, or the interim analysis DCO. An asthma exacerbation was considered severe if it resulted in at least one of the following: use of systemic steroids for at least 3 days, inpatient hospitalization due to asthma or emergency room visit that required systemic steroids, or death due to asthma. The key secondary outcome measure was analyzed at the interim analysis (22 April 2024). Since the key secondary objective was met at the interim analysis, it was not re-tested at final database lock. Since fewer than 50% of participants had an exacerbation event, the median survival time could not be calculated and instead the number of participants with an event is reported.
Time Frame: From treatment initiation until the earliest occurrence of study completion or withdrawal only, regardless of treatment discontinuation, a step-up in maintenance therapy or interim analysis DCO, up to one year following treatment initiation.
Population: Full analysis set; >=12 years
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1209 | 1212
Participants | 64 | 114
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Hazard ratios, 95% confidence intervals for hazard ratios and p-values were estimated using a Cox regression model with treatment group, pre-study asthma therapy, and number of severe exacerbations in the last 12 months prior to randomization as factors. A hazard ratio less than 1 favors the BDA MDI treatment group; Test type: Superiority; p < 0.001, Regression, Cox — The pre-specified alpha (type I error) at the IA was set at 0.003 for the primary and first secondary endpoint; Hazard Ratio (HR) = 0.539, 95% CI 2-sided [0.397 to 0.733]

3. Secondary Outcome: Time to First Severe Asthma Exacerbation, While on Treatment Strategy (Participants Aged >=18 Years)
Description: The time to first severe asthma exacerbation was analyzed under the While on Treatment strategy in the Full analysis set (FAS) and was defined as the length in days from treatment initiation until the date of first severe asthma exacerbation event, including all events that occurred up to the final DCO (20 September 2024). Participants were censored at treatment discontinuation or a step-up in maintenance therapy. An asthma exacerbation was considered severe if it results in at least one of the following: use of systemic steroids for at least 3 days, inpatient hospitalization due to asthma or emergency room visit that required systemic steroids, or death due to asthma. Since fewer than 50% of participants had an exacerbation event, the median survival time could not be calculated and instead the number of participants with an event is reported.
Time Frame: From treatment initiation until the earliest occurrence of study completion, treatment discontinuation or a step-up in maintenance therapy, up to one year following treatment initiation.
Population: Full analysis set; >=18 years
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1180 | 1173
Participants | 71 | 126
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox — The pre-specified type I error for secondary endpoints tested at the final DCO was 0.05. A hierarchical testing strategy was employed to control the two-sided Type I error rate for the secondary endpoints, excluding the first secondary endpoint; Hazard Ratio (HR) = 0.541, 95% CI 2-sided [0.405 to 0.724]

4. Secondary Outcome: Time to First Severe Asthma Exacerbation, Treatment Policy Strategy (Participants Aged >=18 Years)
Description: The time to first severe asthma exacerbation was analyzed under the Treatment Policy strategy in the Full analysis set (FAS) and was defined as the length in days from treatment initiation until the date of first severe asthma exacerbation event, including all events that occurred up to the Final DCO (20 September 2024). Participants were censored at study completion or withdrawal. An asthma exacerbation was considered severe if it resulted in at least one of the following: use of systemic steroids for at least 3 days, inpatient hospitalization due to asthma or emergency room visit that required systemic steroids, or death due to asthma. Since fewer than 50% of participants had an exacerbation event, the median survival time could not be calculated and instead the number of participants with an event is reported.
Time Frame: From treatment initiation until the earliest occurrence of study completion or withdrawal only, regardless of treatment discontinuation or a step-up in maintenance therapy, up to one year following treatment initiation.
Population: Full analysis set; >=18 years
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1180 | 1173
Participants | 73 | 131
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.541, 95% CI 2-sided [0.406 to 0.720]

5. Secondary Outcome: Annualized Severe Asthma Exacerbation Rate, While on Treatment Strategy (Participants Aged >=12 Years)
Description: The annualized exacerbation rate was analyzed under the While on Treatment strategy in the Full analysis set (FAS) and was defined as the length in days from treatment initiation until the date of first severe asthma exacerbation event, including all events that occurred up to the final DCO (20 September 2024). Time at risk was defined as the cumulative number of days in the randomized treatment period across all participants in the treatment group, excluding the days during a severe exacerbation event and the 7 days following it resolving. An asthma exacerbation was considered severe if it resulted in at least one of the following: use of systemic steroids for at least 3 days, inpatient hospitalization due to asthma or emergency room visit that required systemic steroids, or death due to asthma.
Time Frame: as for outcome 3
Population: Full analysis set; >=12 years
Measure: Number (95% Confidence Interval); unit: events per year
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1209 | 1212
events per year | 0.15 [0.11 to 0.20] | 0.32 [0.25 to 0.41]
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Rates, rate ratios and two-sided p-values were estimated from a negative binomial model with treatment, pre-study asthma therapy, and number of severe exacerbations in the last 12 months prior to randomization as factors. A rate ratio less than 1 favors BDA MDI treatment group; Test type: Superiority; p < 0.001, Negative binomial — [p-value comment as in outcome 3, analysis 1]; Rate Ratio = 0.47, 95% CI 2-sided [0.34 to 0.64]

6. Secondary Outcome: Annualized Severe Asthma Exacerbation Rate, While on Treatment Strategy (Participants Aged >=18 Years)
Description: as for outcome 5
Time Frame: as for outcome 3
Population: Full analysis set; >=18 years
Measure: Number (95% Confidence Interval); unit: events per year
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1180 | 1173
events per year | 0.15 [0.12 to 0.20] | 0.33 [0.26 to 0.43]
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Negative binomial — [p-value comment as in outcome 3, analysis 1]; Rate Ratio = 0.46, 95% CI 2-sided [0.33 to 0.63]

7. Secondary Outcome: Total Systemic Glucocorticoid Exposure, While on Treatment Strategy (Participants Aged >=12 Years)
Description: The total systemic glucocorticoid exposure was analyzed under the While on Treatment strategy in the Full analysis set (FAS) and was defined as the cumulative dose of SCS following a severe exacerbation from treatment initiation until study completion, treatment discontinuation or a step-up in maintenance therapy. SCS were normalized to prednisone equivalents when calculating total dose, patients whose total dose could not be normalized are excluded from analysis.
Time Frame: as for outcome 3
Population: Full analysis set; >=12 years
Measure: Mean (Full Range); unit: mg/year
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1204 | 1203
mg/year | 23.2 [0.0 to 2840.8] | 61.9 [0.0 to 21915.0]
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Test type: Superiority; p < 0.001, Wilcoxon rank sum — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Total Systemic Glucocorticoid Exposure, While on Treatment Strategy (Participants Aged >=18 Years)
Description: as for outcome 7
Time Frame: as for outcome 3
Population: Full analysis set; >=18 years
Measure: Mean (Full Range); unit: mg/year
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1175 | 1164
mg/year | 23.0 [0.0 to 2840.8] | 63.0 [0.0 to 21915.0]
Statistical Analysis 1: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Test type: Superiority; p < 0.001, Wilcoxon rank sum — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Total Duration of Systemic Glucocorticoid Exposure, While on Treatment Strategy (Participants Aged >=12 Years)
Description: The total duration of systemic glucocorticoid exposure was analyzed under the While on Treatment strategy in the Full analysis set (FAS) and was defined as the cumulative days of SCS use following a severe exacerbation from treatment initiation until study completion, treatment discontinuation or a step-up in maintenance therapy. SCS were normalized to prednisone equivalents when calculating total dose, patients whose total dose could not be normalized are excluded from analysis.
Time Frame: as for outcome 3
Population: Full analysis set; >=12 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1204 | 1203
days | 0.4 (2.17) | 0.9 (3.66)

10. Secondary Outcome: Total Duration of Systemic Glucocorticoid Exposure, While on Treatment Strategy (Participants Aged >=18 Years)
Description: as for outcome 9
Time Frame: as for outcome 3
Population: Full analysis set; >=18 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
Number analyzed (Participants) | 1175 | 1164
days | 0.4 (2.20) | 0.9 (3.72)

ADVERSE EVENTS:
Time Frame: All-cause mortality (death due to any cause): from randomization up to and including the final DCO (20 September 2024) or study discontinuation, up to 1 year. Treatment-emergent adverse events: from treatment initiation until the earliest occurrence of study completion or treatment discontinuation, up to 1 year.
Description: All-cause mortality was reported for all participants, one reported death occurred post-randomization before first dose of study drug. Adverse events were reported for participants who received at least one dose of study drug, and includes AEs from treatment initiation until the earliest occurrence of study completion or treatment discontinuation.
Arm/Group | BDA MDI (PT027) 160/180 μg | AS MDI (PT007) 180 µg
All-Cause Mortality (participants affected / at risk) | 2/1257 | 1/1259
Serious Adverse Events (participants affected / at risk) | 37/1209 | 37/1212
Other Adverse Events (participants affected / at risk) | 227/1209 | 232/1212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=1209) | AS MDI (PT007) 180 µg (N=1212)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Middle cerebral artery stroke (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Drug screen positive (Investigations) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=1209) | AS MDI (PT007) 180 µg (N=1212)
Upper respiratory tract infection (Infections and infestations) | 65 (74) | 73 (80)
COVID-19 (Infections and infestations) | 62 (63) | 67 (69)
Nasopharyngitis (Infections and infestations) | 45 (46) | 32 (34)
Sinusitis (Infections and infestations) | 38 (41) | 30 (36)
Bronchitis (Infections and infestations) | 29 (30) | 32 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 29 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data or results obtained from this study must not be published without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT05505734/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT05505734/SAP_001.pdf